CLINICAL TRIAL: NCT03893110
Title: Carbon PEEK Versus Titanium Pedicle Screws in the Treatment of Spinal Tumors - A Randomized Controlled Trial
Brief Title: Carbon PEEK Versus Titanium Pedicle Screws in the Treatment of Spinal Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Absence of Co-investigator
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Carbon PEEK
Record Dates: First submitted 2019-02-04; First posted 2019-03-28 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Spinal Tumor
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrumentation with Carbon/PEEK pedicle screw system (Experimental): Posterior instrumentation using a Carbon/PEEK pedicle screw system two levels above and below the affected segment(s). The medical device is a commercial product, bears a conformity marking and is used in accordance with the instructions.
  Interventions: Procedure: surgical stabilization of the spine due to primary and secondary spinal tumors
- Instrumentation with titanium pedicle screw system (Active Comparator): Posterior instrumentation using a titanium pedicle screw system two levels above and below the affected segment(s). The medical device is a commercial product, bears a conformity marking and is used in accordance with the instructions.
  Interventions: Procedure: surgical stabilization of the spine due to primary and secondary spinal tumors

INTERVENTIONS:
Procedure: surgical stabilization of the spine due to primary and secondary spinal tumors — Posterior instrumentation with pedicle screw system

SUMMARY:
Radiation therapy is a cornerstone in the treatment of spinal neoplasms as radical resections are often limited anatomically. Frequently, a surgical stabilization with implants is required. However, metallic implants not only make the CT-based planning of a subsequent radiation therapy more difficult, but might also have an uncontrolled dose modulating effect in adjuvant radiotherapy. At the spine, radiation is limited by the effective dose posed to the relatively radiosensitive spinal cord. While metallic implants might result in an inhomogeneous and uncontrollable dose distribution due to the interface effect, the use of new radiolucent implants consisting of carbon/polyether ether ketone (PEEK) might allow a more homogeneous and predictable dose distribution. This study aims to evaluate the potential benefits of the use of carbon/PEEK pedicle screws during adjuvant radiation therapy and follow-up imaging of spinal tumors.

60 patients will randomized 1:1 into either treatment arm (Pedicle System Carbon/PEEK vs. Pedicle System Titanium). The feasibility of planning the radiation therapy will be evaluated. The postoperatively administered total radiation dose is documented. The radiological visualization of the area of interest will be evaluated The surgical outcome is evaluated by fusion rate, implant integrity and anchorage. Patients will be followed up for 12 months according to local standards.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 99 years of Age
* Primary and secondary spinal tumors of the thoracolumbar spine requiring posterior instrumentation and radiation therapy

Exclusion Criteria:

* Need of cement augmentation or anterior cage support (corpectomy)
* Patients with contraindication against surgical resection
* Patients with incomplete medical records or insufficient imaging

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
radiation dose | within 6 weeks of radiation therapy
  The total radiation dose administered is measured in Gray
feasibility of planning the radiation therapy | before radiation therapy
  evaluated by a subjective score (0-10) stated by an independent radiooncologist using a visual analogue scale from 0 to 10

SECONDARY OUTCOMES:
radiological visualization of the area of interest | during radiation therapy
  evaluated by a subjective score stated by an independent radiologist using a visual analogue scale from 0 to 10
time to recurrence | up to 1 year
  monitoring of recurrence using radiological imaging is performed routinely according to clinical standards

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Farshad, Prof., Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD only available to study personnel. statistical analysis will be done with encoded data only. study results will be published